# Research proposal on evaluation of teen Mental Health First Aid in Hong Kong

by Dr. Benjamin Lai

1 December 2024

Research proposal on evaluation of teen Mental Health First Aid in Hong Kong

Ref: t MHFA 241201p

By Dr. Benjamin Lai

## I. Background information

- 1. Mental health problems in adolescents are on the rise worldwide especially after COVID -19 pandemic. Early detection and intervention should help to reduce the adverse impact of the mental illness on the adolescent. Yet the adolescent may not be able to recognize mental illness, have stigma against the mentally ill and mental health services, and may not seek help even with mental illness. The local situation in Hong Kong has been reviewed and presented in a separate article (Lai, 2024). Teen Mental Health First Aid (t MHFA) is a course developed in Australia for the promotion of mental health literacy including awareness of mental illness, reduction of stigmatizing attitudes towards people with mental illness, and increase in appropriate help-seeking attitude and behavior among adolescents with emerging mental health problems. Mental Health Association of Hong Kong has run the mental health first aid courses in Hong Kong since 2014. The teen MHFA course has been translated and attuned to the local context recently. MHAHK has been funded by the Hong Kong Jockey Club in a two-year project in the development of a quality mental health campus in twenty secondary schools. In the project there will be mental health education programs for teachers, parents and students and mental health promotion activities in the schools. Teen MHFA will be provided to the students in the schools. It is a three-hour course separated into three separate sessions taught by trained instructors of MHAHK.
- 2. The study is an initial evaluation of the t MHFA in secondary school students in Hong Kong. Teen MHFA was initially evaluated in Australia (Hart et al, 2016). The study is a replication of the initial study by Hart et al but followed a quasi-experimental design as in the study of MHFA done in MHAHK (Wong et al, 2015).

3. The study will obtain a baseline information about the awareness of mental illness, the attitude towards the mentally ill and help seeking behavior of secondary school students, and to verify the effectiveness of the teen MHFA course in promotion of mental health literacy of the participants, and to guide the further refinement and development of an effective course. It is hoped that the teen MHFA course can be available to all secondary schools and can help adolescents to develop appropriate mental health literacy at this important phase of development before reaching adulthood.

## II. Study objective:

- 1. To obtain baseline information about the awareness of mental illness, the attitude towards the mentally ill and help seeking behavior of adolescents.
- 2. To evaluate the effectiveness of the teen MHFA course in increasing the awareness of mental illness, facilitating positive change in attitude towards people with mental illness and promoting appropriate help seeking behavior immediately after the course.
- 3. To verify the effectiveness of the teen MHFA course in sustaining its effects after an interval of three months.

# III. Study protocol

## 1. Subjects:

Inclusion criteria:

- 1. Students from mainstream Chinese secondary schools agreeing to host the study
- 2. Studying in Form 4 to Form 6 (About 250 students from different schools)

#### Exclusion criteria:

- 1. Students unable to give consent for the study
- 2. Parents/guardians unable to give consent to the study

#### 2. Control:

- (i) Secondary school students (250 students from the same secondary schools or other secondary schools with similar bandings)
- (ii) Have not attended teen MHFA in the past twelve months

#### 3. Intervention:

All study subjects will be provided with a standard course in the Hong Kong version of Teen MHFA run by trained instructors approved by MHAHK

## 4. Timing of survey

- (i) For subjects: a) Baseline survey is within three weeks before the intervention
  - b) Immediately after the intervention
  - c) Three months after the intervention
- (ii) For control: a) Around the same time of baseline survey for study subjects
  - b) Three months after the baseline survey

# 5. Self-administered questionnaires in survey

- (i) Basic sociodemographic data
- (ii) Mental health literacy (Two vignettes will be provided)
  - (a) Problem recognition
  - (b) Beliefs about help
- (iii) Stigmatizing attitudes
- (iv) Mental health first aid intentions and behaviors
- (v) Mental health status and help seeking status

# 6. Sample size estimation

Given the anticipated effect size of 0.5, a desired statistical power level of 0.8 and a level of .05, it is estimated that a minimum sample size of 128 was needed for a two-group statistical analysis. To cater for the possible inadequate data, the loss to follow up and the wish to have more baseline information about the knowledge, stigma and help seeking attitude of the adolescents a larger size of study subjects is targeted.

- 7. Data analysis
  - (i) Quantitative data are
    - a) digitally entered
    - b) paper questionnaires are employed to facilitate those subjects not able to enter the data digitally
    - c) the data are compiled for basic information about the study subjects and control subjects, and to verify any difference between the study subjects and the control subjects
    - d) the baseline information about awareness of mental illness, the attitude towards the mentally ill and help seeking behavior of adolescents will be compiled
    - e) the null hypothesis will be applied to the statistical analysis in verifying the changes after the intervention in the study subjects
  - (ii) Content analysis of open-ended responses is done by the investigators.
- 8. Ethics: Approval of the study from the research ethics committee of MHAHK
- IV. Adaptation and translation of the questionnaires from Mental Health First Aid International into Chinese will follow the Guidelines for the Process of Cross-Cultural Adaptation of Self-Report Measures (Beaton et al, 2000).

#### References:

Beaton D.E., Bombardier C., Guillemin F., and Ferraz M. B. (2000). Guidelines for the Process of Cross-Cultural Adaptation of Self-Report Measures. SPINE Volume 25, Number 24, pp 3186–3191, 2000

Hart, L.M., Mason, R. J., Kelly, C. M., Cvetkovski, S., and Jorm, A. F. (2016). 'teen Mental Health First Aid': a description of the programme and an initial evaluation. Int J Ment Health Syst,10: 3. Published online 2016 Jan 19. doi: 10.1186/s13033-016-0034-1

Lai B. (2024) Promotion of Mental Health Literacy and Help-Seeking Behaviour of Adolescents with Mental Health Problems - The Local Perspective. Hong Kong Journal of Mental Health 2024, 50(2), 40-49

Wong, D. F.K., Lau, Y., Kwok, S., Wong, P.(2015). Evaluating the effectiveness of mental health first aid programme for Chinese people in Hong Kong. Research on Social Work Practice, 27(1), doi:10.1177/1049731515585149.